CLINICAL TRIAL: NCT01578044
Title: Pilot Intervention to Improve Adherence to Dabigatran for Patients With Atrial Fibillation
Brief Title: Dabigatran Adherence Pilot Intervention for Patients With Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: RRP 11-424
Record Dates: First submitted 2012-04-03; First posted 2012-04-16 (Estimated); Results first posted 2015-06-15 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2018-09

CONDITIONS: Atrial Fibrillation
Keywords: Anti-coagulation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): 1. Patient education: Patients will receive information on dabigatran, including risks, benefits and potential side effects. This information will be re-enforced during the study on a monthly basis during the IVR calls and during the pharmacy service calls to patients.
  2. Tele-monitoring: We will use IVR technology to send patients an automated reminder to refill their dabigatran, rivaroxaban, and apixaban prescriptions. This call will be delivered on day 20 following each dabigatran, rivaroxaban, and apixaban prescription.
  3. Pharmacists follow-up: If dabigatran, rivaroxaban, and apixaban has not been refilled, the pharmacy staff will contact the patient to assess reasons that the patient has not refilled the medication.
  Interventions: Behavioral: Intervention
- Control (Placebo Comparator): Usual care
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Intervention — 1. Patient education: Patients will receive information on dabigatran, including risks, benefits and potential side effects. This information will be re-enforced during the study on a monthly basis during the IVR calls and during the pharmacy service calls to patients.
  2. Tele-monitoring: We will use IVR technology to send patients an automated reminder to refill their dabigatran, rivaroxaban, and apixaban prescriptions. This call will be delivered on day 20 following each dabigatran, rivaroxaban, and apixaban prescriptions.
  3. Pharmacists follow-up: If dabigatran, rivaroxaban, and apixaban have not been refilled, the pharmacy staff will contact the patient to assess reasons that the patient has not refilled the medication.
  Arms: Intervention
Other: Control — Usual care
  Arms: Control

SUMMARY:
Atrial fibrillation is common and increases the risk of clotting especially in patients with multiple clotting risk factors. Patients treated with warfarin, an oral anti-coagulant, require frequent lab monitoring and dose adjustments and are managed in pharmacy staffed anti-coagulation clinics that routinely contact them to remind them about blood draws, re-enforce medication adherence, and adjust dosing based on labs.

Dabigatran, a newly approved medication that may be better for some with atrial fibrillation to lower risk of stroke and clotting, has been found to have fewer drug problems and eliminates lab monitoring need. Following instructions for taking dabigatran is important because it is a twice daily medication requiring monthly refills. Rivaroxaban is a once daily, newly approved Factor Xa inhibitor oral medication, prescribed to reduce risk of stroke and systemic embolism among patients with atrial fibrillation. Apixaban is a twice daily, FDA approved Factor Xa inhibitor oral anticoagulant, prescribed to reduce the risk of stroke and blood clots among patients with atrial fibrillation. In a double-blind RCT, apixaban was found to be superior to warfarin in reducing stroke, systemic embolism, and death. Patients on dabigatran, rivaroxaban, and apixaban will not be followed in anti-coagulation clinics, therefore will not benefit from the support provided by these clinics.

It's anticipated many patients will be switched to dabigatran, rivaroxaban, or apixaban following recent publication of criteria for dabigatran use from the VA National Pharmacy Benefits Management Program, providing an opportune time to conduct the proposed adherence study. We will conduct qualitative interviews with patients(n~30) and pharmacists(n~20) to understand barriers/facilitators to oral anticoagulant adherence. Informed by the findings, we will develop and pilot test a multi faceted intervention to improve adherence among patients recently started on dabigatran/rivaroxaban/apixaban.

Specific study aims:

1. Conduct interviews with a sample of patients (n=30) recently started on dabigatran for atrial fibrillation to determine why patients do or don't take medications
2. Conduct interviews with pharmacists (n=20) in anti-coagulation clinics in order to understand their opinions why patients do or don't take medications
3. Informed by interviews, develop and test an intervention targeting patients/pharmacists to improve adherence to dabigatran/rivaroxaban/apixaban

DETAILED DESCRIPTION:
Hypotheses and Specific Aims: Atrial fibrillation is common and increases the risk of thromboembolic events. Current national guidelines recommend long-term treatment with warfarin, an oral anti-coagulant, for patients with atrial fibrillation and multiple thromboembolic risk factors. Adherence to warfarin is important because of its narrow therapeutic window, which requires frequent lab monitoring (i.e., INR) and dose adjustment. The majority of veterans on warfarin are managed in anti-coagulation clinics staffed by pharmacists who routinely contact patients to remind them to get blood draws, to re-enforce medication adherence, and to adjust warfarin dose based on INR values. Sub-therapeutic anti-coagulation increases the risk of thromboembolic events and is most commonly due to poor medication adherence.

Dabigatran is a newly approved oral factor X inhibitor medication that is more efficacious than warfarin for lowering the risk of stroke and systemic embolism in patients with atrial fibrillation. Additional advantages of dabigatran include fewer drug-drug interactions and standard dosing, eliminating the need for dose titration or lab monitoring. However, adherence is an important consideration with dabigatran because it is a twice a day medication and requires monthly refills due to its formulation, both of which are strong risk factors for non-adherence. In addition, patients taking dabigatran will not be followed in anti-coagulation clinics because there is no lab value to monitor, and therefore, they will no longer benefit from the adherence support provided by these clinics. Non-adherence to chronic cardiovascular medications is common and non-adherence to dabigatran may potentially limit its effectiveness in routine clinical use.

Rivaroxaban is a newly approved, Factor Xa inhibitor, oral medication prescribed to reduce the risk of stroke and systemic embolism among patients with atrial fibrillation. Rivaroxaban is a once daily medication that is recommended to be taken during an evening meal to reduce the potential risk of decreased efficacy of therapy. In a randomized, double-blind study comparing warfarin to Rivaroxaban, Rivaroxaban was found non-inferior to warfarin for the prevention of stroke and systemic embolism in patients with atrial fibrillation, and the risk of major and critically relevant non-major bleeding were similar between the two anticoagulants. In addition, patients taking Rivaroxaban will not be followed in anti-coagulation clinics because there is no lab value to monitor, and therefore, they will no longer benefit from the adherence support provided by these clinics. Non-adherence to chronic cardiovascular medications is common and non-adherence to Rivaroxaban may potentially limit its effectiveness in routine clinical use.

Apixaban is a FDA approved anticoagulant, Factor Xa inhibitor, oral medication prescribed to reduce the risk of stroke and blood clots among patients with atrial fibrillation. Apixaban is taken twice daily. In a double-blind, double-dummy, randomized, non-inferior and superior controlled trial, apixaban was found to be superior to warfarin in reducing stroke, systemic embolism, and death. In addition, patients taking apixaban will not be followed in anti-coagulation clinics because there is no lab value to monitor, and therefore, they will no longer benefit from the adherence support provided by these clinics. Non-adherence to chronic cardiovascular medications is common and non-adherence to apixaban may potentially limit its effectiveness in routine clinical use.

It is anticipated that many patients will be switched to dabigatran following recent publication of criteria for dabigatran use from the VA National Pharmacy Benefits Management Program. This provides an opportune time to conduct the proposed study focusing on adherence to dabigatran, rivaroxaban, and apixaban. We will first perform qualitative interviews with patients (n~30) and pharmacists (n~20) to better understand barriers and facilitators to dabigatran adherence. Informed by the qualitative findings and the literature on interventions to improve cardiovascular medication adherence, we will develop and pilot test a multi-faceted intervention to improve adherence among patients recently started on dabigatran, rivaroxaban, and apixaban.

The proposal is innovative because it proactively addresses dabigatran adherence. This pilot will provide preliminary data for an eventual implementation study to assess the effectiveness of the intervention to improve adherence to dabigatran and patient outcomes, as well as its cost-effectiveness.

Specific aims

1. Conduct in-depth, key informant interviews with a sample of patients (n=30) recently started on dabigatran for atrial fibrillation to determine barriers and facilitators to dabigatran adherence.
2. Conduct in-depth, key informant interviews with a sample of pharmacists (n=20) in anti-coagulation clinics in order to understand their perspectives on barriers and facilitators to patients' maintaining adherence to dabigatran.
3. Informed by the qualitative interviews, develop and pilot test a multi-faceted intervention targeting patients and pharmacists to improve adherence to dabigatran, rivaroxaban, and apixaban.

II. Background and Significance:

Atrial fibrillation is common, affecting 2.2 million Americans and is likely to increase with the aging of the US population. The most devastating sequelae of atrial fibrillation is stroke. National guidelines recommend warfarin, an oral anticoagulant for patients with atrial fibrillation and multiple risk factors (e.g., hypertension, diabetes, older age, stroke or TIA, heart failure) to reduce the stroke risk. Veterans prescribed warfarin are usually managed closely in anti-coagulation clinics. Pharmacists staff these clinics, coordinating blood draws, titrating warfarin dose to maintain therapeutic INR levels, and re-enforcing adherence to therapy. Prior meta-analysis suggests that patients on warfarin managed in these clinics have better anticoagulation control compared to patients followed in non-specialized clinics.

Dabigatran is a newly approved oral direct thrombin inhibitor that was demonstrated to be more efficacious than warfarin for patients with atrial fibrillation. In the RE-LY trial, dabigatran reduced stroke and systemic embolism (Relative risk 0.66; 95% CI, 0.53 to 0.82; P<0.001) with a similar risk of major bleeding (3.36% vs. 3.11% per year; for warfarin vs. dabigatran p=0.31). There are several potential advantages of dabigatran over warfarin, including: 1) standard dosing without need for dose adjustment; 2) no need for lab monitoring; and 3) fewer drug-drug interactions. For these reasons, dabigatran may be preferred by patients requiring chronic anti-coagulation therapy for atrial fibrillation.

Non-adherence to cardiovascular medications is common and limits the effectiveness of medications in routine clinical practice. For most chronic cardiovascular medications, adherence rates begin to decline following the initial prescription, particularly for medications that need to be taken more than once daily, treat asymptomatic conditions and require frequent refills. A prior study found that only ~25% of patient prescribed statins for primary prevention were still adherent at 2 years from the index prescription. The benefits of dabigatran seen in the clinical trial may be significantly lessened if adherence to dabigatran is similar to other chronic cardiovascular medications. This issue of non-adherence is particularly germane to dabigatran because it is a twice a day medication, requires monthly refills due to the formulation of the medication and is used generally as a primary prevention medication for an asymptomatic condition.

In the ROCKET AF Study, Rivaroxaban was found to be non-inferior to warfarin for the prevention of stoke and systemic embolism in patients with atrial fibrillation. Rivaroxaban was non-inferior to warfarin and significantly reduced the risk of stroke or systemic embolism by 21% (hazard ratio (HR), 0.79; 95% confidence interval (CI), 0.66 to 0.96; p less than 0.001). The risk of major and clinically relevant non-major bleeding was similar between both anticoagulant drugs.

In the ARISTOTLE trial, apixaban had a greater reduction of hemorrhagic stroke compared to the warfarin group (HR 0.51; 95% CI 0.35 to 0.75; p less than 0.001). For the secondary outcome of death from any cause, apixaban was superior to warfarin (HR 0.89; 95% CL 0.8 to 0.998; p=0.047).

Pharmacists have helped patients to improve adherence to cardiovascular medications and intermediate outcomes such as BP and LDL control. For anticoagulation therapy, pharmacists have helped patients maintain better INR control via anti-coagulation clinics compared to patients not managed in these clinics. Specific components of anti-coagulation clinics that have been found to be particularly helpful for improving adherence include computerized patient monitoring that identifies delinquent patients (i.e., for lab monitoring) and frequent contacts with the patient. An intervention focusing on adherence involving pharmacists can have the potential to improve dabigatran, rivaroxaban, and apixaban use so that the benefits demonstrated in the clinical trials for dabigatran can be realized in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have transitioned from warfarin to dabigatran, rivaroxaban, or apixaban or are recently started on anti-coagulation for atrial fibrillation with dabigatran, rivaroxaban, or apixaban will be eligible to be interviewed and partake in the intervention.
* Pharmacists from the Denver VA Medical Center and who work in the anti-coagulation clinics will be eligible to be interviewed.

Exclusion Criteria:

* Patients who prefer a telephone interview but do not have a telephone or cell phone will be excluded.
* Patients for whom the VA is not the primary source of care will also be excluded.
* Pregnant patients will be excluded.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Ho, MD PhD, Principal Investigator — VA Eastern Colorado Health Care System, Denver, CO
Locations (1):
- VA Eastern Colorado Health Care System, Denver, CO, Denver, Colorado, United States

REFERENCES:
- [Result] Shore S, Carey EP, Turakhia MP, Jackevicius CA, Cunningham F, Pilote L, Bradley SM, Maddox TM, Grunwald GK, Baron AE, Rumsfeld JS, Varosy PD, Schneider PM, Marzec LN, Ho PM. Adherence to dabigatran therapy and longitudinal patient outcomes: insights from the veterans health administration. Am Heart J. 2014 Jun;167(6):810-7. doi: 10.1016/j.ahj.2014.03.023. Epub 2014 Apr 5. PMID 24890529
- [Result] Shore S, Carey E, Turakhia M, Jackevicius CA, Cunningham F, Pilote L, Baron A, Grunwald G, Bradley SM, Maddox TM, Rumsfeld JS, Varosy PD, Ho M. Patterns of Adherence to Dabigatran and its Association with Outcomes. [Abstract]. Circulation. 2013 Nov 26; 128(22 Suppl):A16864.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who are new starts on dabigatran, apixaban, and rivaroxaban and have completed the initial 3-month pharmacy follow-up will be approached by a pharmacist to inquire about their interest in participating in our study. Patients interested will verbally consent to participate and will then be randomized to the intervention or control group.
Groups:
- Intervention Group: Intervention patients will receive the following:
  1. Patient education: All patients will receive information on their oral anticoagulant, including risks, benefits, and potential side effects. Intervention patients will receive additional materials at the beginning of the study through the mail.
  2. Tele-monitoring: IVR technology will be used to send patients automated reminders to refill their dabigatran, rivaroxaban, and apixaban prescriptions. This call will be delivered on day 20 following each anticoagulant prescription.
  3. Pharmacists follow-up: If dabigatran, rivaroxaban, and apixaban has not been refilled, the pharmacy staff will contact the patient to assess reasons that the patient has not refilled the medication.
- Usual Care: Usual care patients will receive information on dabigatran, apixaban, and rivaroxaban including risks, benefits and potential side effects.
  Following the end of the study, the usual care patients will receive the additional educational materials the intervention group received during the study.
Period: Overall Study
Arm/Group | Intervention Group | Usual Care
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intervention Group: Patients who are randomized to the intervention group will receive the following:
  1. Patient education: Patients will receive information on dabigatran, apixaban, and rivaroxaban, including risks, benefits and potential side effects. This information will be re-enforced during the study on a monthly basis during the IVR calls and during the pharmacy service calls to patients.
  2. Tele-monitoring: IVR technology will be used to send patients automated reminders to refill their dabigatran, rivaroxaban, and apixaban prescriptions. This call will be delivered on day 20 following each anticoagulant prescription.
  3. Pharmacy follow-up: If the anticoagulant has not been refilled, the pharmacy staff will contact the patient to assess reasons the patient has not refilled the medication.
- Usual Care Group: Usual care
  Usual care patients will receive information on dabigatran, apixaban, and rivaroxaban including risks, benefits and potential side effects.
  Following the end of the study, the usual care patients will receive the additional educational materials the intervention group received during the study.
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Usual Care Group | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 6 | 6 | 12
Age, Continuous [Mean (Full Range); unit: Years] | 70.5 [67 to 78] | 69.3 [63 to 84] | 69.9 [63 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 6 | 12
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Gaps Days Between Prescription Refills for Dabigatran, Rivaroxaban, and Apixaban
Description: The investigators will calculate the # of gap days between refills for dabigatran/rivaroxaban/apixaban for each3 and 6 months of the pilot intervention. This will be based on pharmacy refill data and calculated using the date dabigatran/rivaroxaban/apixaban was dispensed and the # of days supplied for that prescription. We will add the # of gap days for each 3 and 6 months of the pilot for each patient, and compare the total # of gaps days between intervention and usual care patients. The gap days between refills is a validated measure of adherence and identifies patients with sub-optimal adherence.A negative gap day value indicates that participants received the refill prior to completion of the previous prescription.
Time Frame: 3 and 6 months
Measure: Number; unit: days
Groups:
- Intervention Group: 1. Patient education: Patients will receive information on dabigatran, including risks, benefits and potential side effects. This information will be re-enforced during the study on a monthly basis during the IVR calls and during the pharmacy service calls to patients.
  2. Tele-monitoring: We will use IVR technology to send patients an automated reminder to refill their dabigatran, rivaroxaban, and apixaban prescriptions. This call will be delivered on day 20 following each dabigatran, rivaroxaban, and apixaban prescription.
  3. Pharmacists follow-up: If dabigatran, rivaroxaban, and apixaban has not been refilled, the pharmacy staff will contact the patient to assess reasons that the patient has not refilled the medication.
- Usual Care Group: All usual care patients will receive information on dabigatran, rivaroxaban, and apixaban, including risks, benefits, and potential side effects. Additionally, following their time in the study, the usual care patients will receive the additional educational materials the usual care received.
Arm/Group | Intervention Group | Usual Care Group
Number analyzed (Participants) | 6 | 6
days
  # of Patient gap days for 3-months of intervention | 43 | 51
  # of Patient gap days for 6-months of intervention | 41 | -5

ADVERSE EVENTS:
Groups:
- Usual Care Group: Usual care
  All patients will receive information on dabigatran, rivaroxaban, and apixaban, including risks, benefits, and potential side effects. Also, following their enrollment in the study will receive the additional educational materials given to the intervention group during their time in the study.
Arm/Group | Intervention Group | Usual Care Group
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes